CLINICAL TRIAL: NCT02929251
Title: Multicentre, Randomized, Multi-arm Trial Comparing the Efficacy and Safety of Adalimumab, Anakinra and Tocilizumab in Subjects With Non-infectious Refractory Uveitis RUBI: Refractory Uveitis BIotherapies
Brief Title: Randomized Trial Comparing Efficacy of Adalimumab, Anakinra and Tocilizumab in Non-infectious Refractory Uveitis
Acronym: RUBI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P150945; 2016-002284-34 (EudraCT Number)
Record Dates: First submitted 2016-10-07; First posted 2016-10-11 (Estimated); Last update posted 2025-09-16 (Actual); Status verified 2024-06

CONDITIONS: Uveitis; Biotherapy
MeSH Terms: conditions — Uveitis | interventions — Interleukin 1 Receptor Antagonist Protein; tocilizumab; Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Adalimumab (Active Comparator): Adalimumab (40mg/14 days subcutaneously) (n=40) for 16 weeks
  Interventions: Drug: Adalimumab
- Anakinra (Experimental): Anakinra (100 mg/day subcutaneously) (n=40) for 16 weeks
  Interventions: Drug: Anakinra
- Tocilizumab (Experimental): Tocilizumab (162 mg/7 days subcutaneously) (n=40) for 16 weeks.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Anakinra — Anakinra (100 mg/day subcutaneously) (n=40) for 16 weeks
  Arms: Anakinra
Drug: Tocilizumab — Tocilizumab (162 mg/7 days subcutaneously) (n=40) for 16 weeks.
  Arms: Tocilizumab
Drug: Adalimumab — Adalimumab (40mg/14 days subcutaneously) (n=40) for 16 weeks
  Arms: Adalimumab

SUMMARY:
RUBI, is the first prospective randomized, head to head study, comparing Adalimumab to either anakinra, or tocilizumab in refractory Non Infectious Uveitis (NIU). There is no firm evidence or randomized controlled trials directly addressing the best biologic agent in severe and refractory NIU. NIU can cause devastating visual loss and up to 20% of legal blindness. Corticosteroids and immunosuppressants failed to demonstrate sustainable remission over 70 % of refractory/relapsing severe uveitis. The incidence of blindness in NIU has been dramatically reduced in the recent years with the use of biologics, raising the question of whether these compounds should be used earlier in the treatment of severe non infectious uveitis. Contrasting with immunosuppressors, biotherapies act rapidly and are highly effective in steroid's sparing thus preventing occurrence of cataract and/or glaucoma.

Despite a strong rationale, these compounds are not yet approved in uveitis, which guarantees the innovative nature of this study that aims selecting or dropping any arm when evidence of efficacy already exists.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written, informed consent prior to the performance of any study specific procedures
2. Diagnosis of non-infectious intermediate, posterior-, or pan-uveitis in at least one eye fulfilling the International Study Group Classification Criteria (Standardization of Uveitis Nomenclature [SUN] criteria) of posterior, or pan- uveitis confirmed by documented medical history
3. Currently uncontrolled uveitic disease. Uncontrolled uveitic disease is defined as fulfilling one of the two following criteria at Inclusion:

   * Active inflammatory chorioretinal and/or inflammatory retinal vascular lesions and/or macular edema (CRT ≥300 microns) OR
   * Vitreous haze grade ≥4 on the Miami 9-step scale (or VH >1+ according to SUN/NEI classification)
4. a. Patient who are receiving prednisone ≥10 mg/day and <80mg/day (or equivalent dose of another corticosteroid) at stable dose 30 days prior to the first study drug administration on Day 0 and who received at least 1 other systemic immunosuppressant (All systemic immunosuppressants must have been discontinued 30 days prior to the first study drug administration on Day 0), or, b. Patient who received IFN alpha (All systemic immunosuppressants must have been discontinued 30 days prior to the first study drug administration on Day 0), or, c. To be intolerant to immunosuppressant
5. Best corrected visual acuity (BCVA) by ETDRS ≥ to 20/400 in either eye
6. Stable dose for two weeks prior to inclusion of topical corticosteroids and/or NSAIDs
7. Male or female , Age >= 18 years at Inclusion
8. Weight 40 - 120 kg (88.2 - 264 lbs) at Inclusion
9. Chest X-ray or thoracic CT scan results (postero-anterior and lateral) within 12 weeks prior to Inclusion with no evidence of active Tuberculosis, active infection, or malignancy
10. For female subjects of child-bearing age, a negative serum or urine pregnancy test
11. For subjects with reproductive potential, a willingness to use contraceptive measures adequate to prevent the subject or the subject's partner from becoming pregnant during the study and 3 and 5 months after stopping therapy for roactemra and adalimumab, respectively. Birth control methods which may be considered as highly effective methods that can achieve a failure rate of less than 1% per year when used consistently and correctly are considered as highly effective birth control methods (according to CTFG recommendations). Such methods include :

    * combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation 1:

      * oral
      * intravaginal
      * transdermal
    * progestogen-only hormonal contraception associated with inhibition of ovulation 1:

      * oral
      * injectable
      * implantable
    * intrauterine device (IUD)
    * intrauterine hormone-releasing system ( IUS)
    * bilateral tubal occlusion
    * vasectomised partner
    * sexual abstinence (In the context of this guidance sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject).
12. A QuantiFERON®-Tuberculosis (TB) test within 6 months prior to Screening

Exclusion Criteria:

1. Infectious uveitis, masquerade syndromes (idiopathic uveitis is permitted)
2. Isolated anterior uveitis
3. Presence of cataract or posterior capsular opacification so severe that an assessment of the posterior segment of either eye is inadequate or impossible
4. Contraindication to mydriasis in either eye or presence of posterior synechiae in the study eye such that mydriasis is inadequate for posterior segment examination
5. Intraocular pressure ≥ 25 mmHg by Goldmann tonometry or advanced glaucoma in either eye
6. Monocular patient
7. Active tuberculosis
8. Known positive syphilis serology, HIV antibody, hepatitis B surface antigen and/or anti-nucleocapsid antibody of hepatitis B virus and/or Hepatitis C virus, within 1 month prior to inclusion.
9. History of malignancy within 5 years prior to Inclusion other than carcinoma in situ of the cervix or adequately treated, non-metastatic squamous or basal cell carcinoma of the skin.
10. History of severe allergic or anaphylactic reactions to monoclonal antibodies
11. Infectious disease:

    * Fever or infection requiring treatment with antibiotics within 3 weeks prior to Inclusion
    * History of recurrent infection or predisposition to infection
12. Known immunodeficiency
13. History of multiple sclerosis and/or demyelinating disorder
14. Laboratory values assessed during Inclusion:

    * Hemoglobin < 8g/dL
    * White Blood Cell Count (WBC) < 2.0 x 10^3/mm3
    * Platelet count < 80 x 10^3/mm3
    * Glomerular filtration rates (GFR) <30ml/min.
    * Transaminases > 3 times upper normal value
15. Use of the following systemic treatments during the specified periods:

    * Any other previous systemic biologic therapy
    * Treatment with any systemic alkylating agents within 12 months prior to Inclusion or between Inclusion and Day 0 (e.g., cyclophosphamide, chlorambucil)
    * Any live (attenuated) vaccine within 3 months prior to Inclusion
16. Use of the following ocular treatments during the specified periods:

    * Previous anti Vascular Endothelial Growth Factor (VEGF) intravitreal therapy (applied to both eyes) within 3 months prior to Inclusion, or anticipated use during the study period
    * Treatment with dexamethasone intravitreal implant [Ozurdex®]) within 6 months prior to Inclusion
    * Intravitreal corticosteroids within 3 months prior to Inclusion. Previous Subtenon's corticosteroid injections are permitted if administered at least 2 months prior to Inclusion
17. Stage III and IV New York Heart Association (NYHA) cardiac insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2022-01-29 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with at least 2-step reduction in Vitreous Haze (according to Miami 9-step Scale) and with a dose <= 0.1 mg/Kg/day of prednisone (or equivalent oral corticosteroid) | Week 16
  Percentage of patients with at least 2-step reduction in Vitreous Haze (according to Miami 9-step Scale) and with a dose <= 0.1 mg/Kg/day of prednisone (or equivalent oral corticosteroid)

SECONDARY OUTCOMES:
Mean change from baseline in Vitreous Haze | Week 4, 8, 12, 16, 24
  Mean change from baseline in Vitreous Haze
Percentage of patients with anterior chamber score = 0 or at least 2-step reduction in score (Tyndall and flare according to the Standardization of Uveitis Nomenclature (SUN) classification) | Week 4, 8, 12, 16, 24
Mean change from baseline in BCVA (ETDRS letters score) | Week 4, 8, 12, 16, 24
Mean change from baseline in central retinal thickness measured with Optical Coherence Tomography (OCT) | Week 4, 8, 12, 16, 24
Percentage of patients with Central Retinal Thickness (CRT) <300 microns | Week 4, 8, 12, 16, 24
Percentage of patients without retinal vessel leakage on fluorescein angiography | Week 4, 8, 12, 16, 24
Percent meeting targets ≤ 0.1 mg/day prednisone | week 16
Mean change in prednisone dose | Week 4, 8, 12, 16, 24
Mean dose of prednisone | week 16
Cumulative dose of prednisone | week 16
Time to response onset | week 16
Time to relapse of uveitis | week 30
Number of relapse of uveitis | week 30
Underlying systemic disease | week 4, 8, 12, 16, 24
  Complete remission of extra opthalmologic sign of Behcet disease or sarcoidosis
Percentage of adverse event | week 4, 8, 12, 16, 24
Percentage of serious adverse event | week 4, 8, 12, 16, 24
time to treatment failure | week 30

CONTACTS AND LOCATIONS:
Overall Officials: David Saadoun, MD PHD, Principal Investigator — APHP
Locations (27):
- France (27):
  - Hopital la pitié salpetriere - Médecine interne 1, Paris, paris
  - Hopital Avicenne - CRC, Bobigny
  - Hopital Avicenne - Ophtalmologie, Bobigny
  - Hopital Avicenne- Médecine interne, Bobigny
  - Hopital Pellegrin, Bordeaux
  - Hopital Saint André - Médecine interne, Bordeaux
  - CHU Clermont-Ferrand - Hopital Gabriel Montpied - Médecine interne, Clermont-Ferrand
  - CHU Clermont-Ferrand - Hopital Gabriel Montpied - Ophtalmologie, Clermont-Ferrand
  - CHU Dijon Bourgogne -Ophtalmologie, Dijon
  - CHU Dijon Bourgogne Médecine Interne et Maladies Systémiques - Médecine 2 / SOC 2, Dijon
  - HCL - Hôpital de la Croix Rousse - Médecine interne, Lyon
  - HCL - Hôpital de la Croix Rousse - Ophtalmologie, Lyon
  - CHRU de Nancy - Médecine interne, Nancy
  - CHRU de Nancy, Nancy
  - CHNO des Quinze Vingt - Médecine interne, Paris
  - CHNO des Quinze Vingt - Ophtalmologie, Paris
  - CHNO des Quinze Vingt, Paris
  - Hopital Pitié Salpetriere, Paris
  - Hopital Rotchild - Médecine interne, Paris
  - Hopital Rotchild - Ophtalmologie, Paris
  - Hôpital de la pitié salpêtrière - Ophtalmologie, Paris
  - CHRU de Rennes Hopital Sud Médecine interne, Rennes
  - CHU Rennes - Hopital Ponchaillou - Ophtalmologie, Rennes
  - CHU Rouen - Hopital Charles Nicolle - Ophtalmologie, Rouen
  - CHU Rouen - Hopital Charles Nicolle - Médecine interne, Rougé
  - CHU TOULOUSE - HOPITAL PIERRE PAUL RIQUET - Ophtalmologie, Toulouse
  - CHU Toulouse - Hopital Rangueil, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saadoun D, Ghembaza A, Touhami S, Girszyn N, Bielefeld P, Seve P, Pugnet G, Andre M, Leclercq M, Rogier T, Ribeiro E, Hie M, Clavel G, Abad S, Stanescu-Segall D, Toutee A, Gueudry J, Bron A, Kodjikian L, Soler V, Chiambaretta F, Sene T, Titah SMC, Heron E, Moulana A, Trad S, Terrada C, Massamba N, Raked N, Resche-Rigon M, Domont F, Desbois AC, Maalouf G, Vautier M, Cacoub P, Desseaux K, Vieira M, Biard L, Bodaghi B. Adalimumab, Anakinra and Tocilizumab in patients with non-infectious Uveitis: A multicenter randomized controlled trial. Am J Ophthalmol. 2026 Feb 3:S0002-9394(26)00052-8. doi: 10.1016/j.ajo.2026.01.037. Online ahead of print. PMID 41643758